CLINICAL TRIAL: NCT03570775
Title: Effectiveness, Safety and Perceptions With the Use of One Phototherapy LED Device: a Sleeping Bag for Hospital Treatment of Neonatal Jaundice
Brief Title: Effectiveness, Safety and Perceptions With the Use of One LED Sleeping Bag Device in the Treatment of Neonatal Jaundice
Acronym: LEDlightT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathalie Charpak (Other)
Collaborators: Hospital Universitario San Ignacio (Other); Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor-Investigator, Nathalie Charpak, Director, Kangaroo Foundation
Organization: Kangaroo Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/186
Record Dates: First submitted 2018-06-04; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Phototherapy; Jaundice, Neonatal
Keywords: hyperbilirubinemia; treatment; devices; newborn; phototherapy
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial with newborns over 2000 grams of birth weight and diagnosis of indirect hyperbilirubinemia, requiring phototherapy. Patients were randomized to phototherapy with the LED sleeping bag or conventional phototherapy with blue light panels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Neomedlight" Sleeping bag phototherapy (Experimental): Phototherapy device with LED light + fiber optic mesh
  Interventions: Device: Sleeping bag phototherapy
- Conventional phototherapy (Active Comparator): LU-6T model: phototherapy device with six fluorescent tubes, four white and two blue, with adjustment of inclination and height incorporated.
  Interventions: Device: Conventional phototherapy

INTERVENTIONS:
Device: Sleeping bag phototherapy — This device has a LED light emitter that incorporates one fiber optic mesh and is protected by a vinyl cover and a disposable liner for patient comfort and hygiene. The phototherapy sleeping bag is conceived with the aim of increasing the surface of phototherapy by means of a double exposure: ventral and dorsal, which allows the insertion of two phototherapy devices of 20x30 centimeters. The ventral and dorsal caps incorporate mesh optical fibers that are connected to the light emitter, in which the phototherapy time can be programmed. The fiber optic meshes are protected by a vinyl cover and a disposable lining for patient comfort and hygiene.
  Other Names: "Neomedlight" sleeping bag phototherapy device
  Arms: "Neomedlight" Sleeping bag phototherapy
Device: Conventional phototherapy — This is a phototherapy device with six fluorescent tubes, four white and two blue, with adjustment of inclination and height incorporated. The device has a minimum height of 106 cm and a maximum of 152 cm, a depth of 64 cm and a width of 72 cm. The manufacturer recommends not using the lamp at distances of less than 50 cm because, although the heat radiation is minimal, this can influence distances less than 50 cm when the child is also exposed to infrared thermal radiation, typical of the servo cribs It is recommended to control temperature and eye protection due to the risk of ophthalmic injury from light, since the intensity of the light is concentrated in a single point.
  Other Names: LU-6T phototherapy
  Arms: Conventional phototherapy

SUMMARY:
Objective: to evaluate the effectiveness, safety and level of satisfaction of parents and healthcare team with one innovative device for phototherapy to which a LED light mesh has been incorporated(a sleeping bag), comparing it with conventional hospital phototherapy. Methods: randomized controlled clinical trial with newborns more than 2000 g of birth weight hospitalized requiring phototherapy. The study protocol was evaluated and accepted by the San Ignacio Hospital and "Pontificia Universidad Javeriana" research committee. Informed consent was requested from parents and the authors declared no conflict of interest. Sample size and allocation: using the STATA 12 program, a sample size of 58 patients was calculated, 29 for each group, with significance level of 0.05, power of 80% and difference in bilirubin decreasing of at least 0,1 mg/dl/h with standard deviation of 0.14 mg/dl/h. A computer program randomized the allocation to the intervention and the concealment of the assignment was through sealed opaque envelopes. Bilirubin levels were taken at the start of phototherapy. Controls were at the beginning, every 8 hours and every 12 hours at the time of bilirubin stabilization in the case of hemolysis, or every 24 hours depending on risk factors. Axillary temperature was measured at the beginning of phototherapy, at 30 min, 60 min, 120 min and every 24 hours during intervention. Physical examination and daily water balance were performed. Parents and health personnel answered a survey on comfort and perceptions with the use of the devices at the end of phototherapy. Analysis: Comparison of means was made for the decrease of bilirubin levels and body temperatures and chi-square for incidence of side effects and results of the survey.

DETAILED DESCRIPTION:
Background: Jaundice due to hyperbilirubinemia is the most common entity that requires medical management in neonates. About 50% of full-term newborns and 80% of premature infants develop jaundice. The effectiveness of phototherapy for neonatal jaundice depends on two factors: the spectrum of light emitted and the spectral irradiation of light. An ideal phototherapy device should have a broad light emission surface, in order to cover the maximum of the body surface in the horizontal plane, it should be durable, generate relatively little heat and provide a wavelength and light intensity (radiation) optimal (460-490nm and ≥ 30uw / cm2 / nm). The conventional phototherapy devices use fluorescent lamps that emit heat and require eye protectors, in addition to increasing water losses, which requires a permanent monitoring of vital functions and temperature. Its use imposes hospitalization and consequently mother-child separation, always traumatic. The most recent devices use light emitting diodes (LED light) as the light source. Objective: to evaluate the effectiveness, safety and level of satisfaction of parents and healthcare team with one innovative device for phototherapy to which a LED light mesh has been incorporated (a sleeping bag ), comparing it with conventional phototherapy for hospitalized patients. Methods: randomized controlled clinical trial with newborns more than 2000 g of birth weight that required phototherapy according to the guidelines of the American Academy of Pediatrics, admitted to the "Hospital Universitario San Ignacio Neonata Care Unit (NCU)" . The Protocol was evaluated and accepted by the Hospital and "Pontificia Universidad Javeriana" research committee. Informed consent was requested from parents and the authors declared no conflict of interest. Sample size and allocation: using the STATA 12 program, a sample size of 58 patients was calculated, 29 for each group, with significance level of 0.05, power of 80% and difference in bilirubin decreasing of at least 0,1 mg/dl/h with standard deviation of 0.14 mg/dl/h. A computer program randomized the allocation to the intervention and the concealment of the assignment was through sealed opaque envelopes. Seric bilirubin levels were taken at the start and at the end of phototherapy. Controls were at the beginning, every 8 hours and every 12 hours at the time of bilirubin stabilization in the case of hemolysis, or every 24 hours depending on risk factors. Axillary temperature was measured at the beginning and during phototherapy. Physical examination and daily water balance were performed. Parents and health personnel answered a survey on comfort and perceptions with the use of the devices at the end of the intervention. Analysis: Comparison of means was made for decrease of bilirubin levels and body temperatures and chi-square for incidence of side effects and results of the survey.

ELIGIBILITY:
Inclusion Criteria:

* Hyperbilirubinemia requiring phototherapy according to the guidelines of the American Academy of Pediatrics and management recommendations for preterm infants under 35 weeks, adopted by the newborn unit of San Ignacio University Hospital.
* Birth weight more than 2000 grams.
* Parents are required to sign informed consent where they agree to participate in the study

Exclusion Criteria:

* Diagnosis of pemphigus, scalded skin or burns that make phototherapy difficult.
* Patient who requires transfer for management in another institution by their health insurer.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Bilirubin reduction rate in mg/dl/h | through study completion, an average of 5 days
  Bilirubin lowering rate (initial seric bilirubin- final seric bilirubin/time of phototherapy)

SECONDARY OUTCOMES:
Patient temperature during phototherapy | through study completion, an average of 5 days
  Axillary temperatures at 30 min, 60 min, 120 min, diary and at the end of phototherapy
Incidence of skin lesions related to phototherapy | through study completion, an average of 5 days
  rash, burns, etc... related to phototherapy
Incidence of dehydration related to phototherapy | through study completion, an average of 5 days
  documented with water balance and weight
Incidence of diarrhea related to phototherapy | through study completion, an average of 5 days
  documented diarrhea
Incidence of other side effects related to phototherapy | through study completion, an average of 5 days
  other effects recorded in clinic history related to phototherapy
Perceptions of parents with the use of devices (comfort, heat, humidity, ease of breastfeeding, proximity and possibility of contact with the baby) | at study completion, an average of 5 days
  Validated survey at the end of treatment with Likert Scale( range 1 to 7. 1= completely uncomfortable. 7= completely comfortable. 4=indifferent)
Perceptions of the health team with the use of the devices (comfort, heat, humidity, ease of breastfeeding, proximity and possibility of contact with the baby) | at study completion, an average of 5 days
  Validated survey at the end of treatment with Likert Scale( range 1 to 7. 1= completely uncomfortable. 7= completely comfortable. 4=indifferent)
Incidence of mortality | through study completion, an average of 5 days
  Mortality related to treatment
Incidence of exchange transfusion | through study completion, an average of 5 days
  Incidence of patients who required exchange transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Andrade, Dr., Study Chair — Hospital Universitario San Ignacio; Nathalie Charpak, Dr., Study Director — Kangaroo Foundation
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No